CLINICAL TRIAL: NCT01207323
Title: A Phase I, Open-Label, Dose-Escalation Study of the Safety and Pharmacokinetics of MEHD7945A Administered Intravenously to Patients With Locally Advanced or Metastatic Epithelial Tumors
Brief Title: A Study of the Safety and Pharmacokinetics (PK) of MEHD7945A in Participants With Locally Advanced or Metastatic Epithelial Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAF4873g; GO00765 (Other: Genentech, Inc.); 2010-022217-26 (EudraCT Number)
Record Dates: First submitted 2010-09-20; First posted 2010-09-22 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Epithelial Tumors, Malignant
MeSH Terms: conditions — Carcinoma | interventions — MEHD7945A

ARMS (2):
- Dose Escalation (MEHD7945A) (Experimental): Participants will receive intravenous (IV) infusion of MEHD7945A in escalating doses Q2W until MTD is reached or up to disease progression as determined by the investigator, intolerable toxicity, withdrawal of consent, or death, whichever occurs first. Approximately 5 dose levels between 1 and 30 mg/kg will be evaluated.
  Interventions: Drug: MEHD7945A
- Dose Expansion (MEHD7945A) (Experimental): Participants will receive IV infusion of MEHD7945A Q2W at or below the MTD (decided from dose escalation part) up to disease progression as determined by the investigator, intolerable toxicity, withdrawal of consent, or death, whichever occurs first.
  Interventions: Drug: MEHD7945A

INTERVENTIONS:
Drug: MEHD7945A — MEHD7945A will be administered as specified in the individual arms.

SUMMARY:
This is a Phase I, multicenter, open-label study of MEHD7945A in participants with incurable, locally advanced, or metastatic epithelial malignancies that have progressed despite standard therapy or for which no standard therapy exists. The study will be conducted in two stages: a dose escalation stage and an expansion stage. The dose-escalation stage is designed to evaluate the safety, tolerability, and PK of MEHD7945A administered (at five dose levels from 1 to 30 milligrams per kilogram [mg/kg]) every 2 week (Q2W). An expansion stage will be initiated after establishment of maximum tolerated dose (MTD) in dose escalation stage. Participants with refractory or recurrent metastatic colorectal cancer (CRC), non-small cell lung cancer (NSCLC), head and neck squamous cell carcinoma (HNSCC), and pancreatic cancer will be enrolled in an expansion stage to better characterize the safety, tolerability, PK and preliminary assessment of the anti-tumor activity of MEHD7945A.

ELIGIBILITY:
Inclusion Criteria:

* Life expectancy greater than or equal to (>/=) 12 weeks
* Availability and willingness to provide sufficient tumor tissue sample for testing
* Dose-escalation stage: Participants with histologically documented incurable, locally advanced, or metastatic epithelial malignancy that has progressed despite standard therapy or for which no standard therapy exists
* Expansion stage: Participants with one of the following epithelial, histologically-documented, incurable, locally advanced, or metastatic tumor that has progressed despite standard therapy or for which no standard therapy exists: CRC, NSCLC, HNSCC, or pancreatic cancer
* Use of an effective means of contraception (e.g., abstinence, hormonal or double barrier method, surgically sterilized partner) for men and women of childbearing potential while enrolled in the study

Exclusion Criteria:

* Less than (<) 4 weeks since the last anti-tumor therapy prior to Day 1 of study treatment
* Major surgical procedure within 4 weeks prior to Cycle 1, Day 1
* Leptomeningeal disease as the only manifestation of the current malignancy
* Active infection requiring IV antibiotics
* Active autoimmune disease that is not controlled by nonsteroidal anti-inflammatory drugs
* Symptomatic hypercalcemia requiring continued use of bisphosphonate therapy
* Current severe, uncontrolled systemic disease
* History of cardiac heart failure of any New York Heart Association criteria or serious cardiac arrhythmia requiring treatment
* History of myocardial infarction within 6 months before Cycle 1, Day 1, or history of unstable angina
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* History of interstitial lung disease
* History of severe allergic or hypersensitivity reaction to other therapeutic antibodies that required discontinuation of therapy
* Known human immunodeficiency virus (HIV) infection
* Primary central nervous system (CNS) malignancy or untreated/active CNS metastases
* Significant traumatic injury within 4 weeks before Cycle 1, Day 1
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2010-11-09 (Actual); Primary Completion 2013-12-03 (Actual); Study Completion 2018-04-23 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Dose-Limiting Toxicities (DLTs) of MEHD7945A | Days 1-28
Maximum Tolerated Dose (MTD) of MEHD7945A | Days 1-28
Percentage of Participants With Adverse Events | Baseline up to approximately 6.75 years
Percentage of Participants With Anti-MEHD7945A Antibodies | Baseline up to approximately 6.75 years (assessed at predose [0 to 4 hours {Hr}] on Day 1 [D1] of Cycles [Cy] 1, 2, 4 [1 Cycle: 14 days], at the study completion/early termination (ET) visit [up to approximately 6.75 years])

SECONDARY OUTCOMES:
Area Under the Concentration-Time Curve (AUC) of MEHD7945A | Predose (0-4 Hr), 0.5, 4, 24, 72Hr post Cy1 D1 dose (infusion duration=1.5 Hr); Day 8 of Cy 1, 2, 4; predose, 0.5 Hr postose on Day 1 of Cy2, 3, 4, 6, every 4 Cy thereafter (up to Cy16); study completion/ET (approximately 6.75 years) (Cy=14 days)
Maximum Serum Concentration (Cmax) of MEHD7945A | Predose (0-4 Hr), 0.5, 4, 24, 72Hr post Cy1 D1 dose (infusion duration=1.5 Hr); Day 8 of Cy 1, 2, 4; predose, 0.5 Hr postose on Day 1 of Cy2, 3, 4, 6, every 4 Cy thereafter (up to Cy16); study completion/ET (approximately 6.75 years) (Cy=14 days)
Minimum (Trough) Concentration (Cmin) of MEHD7945A | Predose (0 to 4 hours) on D1 of Cy1,2,3,4,6, every 4 Cy thereafter (up to Cy16 ); study completion/ET (up to approximately 6.75 years) (Cy=14 days)
Clearance (Cl) of MEHD7945A | Predose (0-4 Hr), 0.5, 4, 24, 72Hr post Cy1 D1 dose (infusion duration=1.5 Hr); Day 8 of Cy 1, 2, 4; predose, 0.5 Hr postose on Day 1 of Cy2, 3, 4, 6, every 4 Cy thereafter (up to Cy16); study completion/ET (approximately 6.75 years) (Cy=14 days)
Volume of Distribution at Steady State (Vss) of MEHD7945A | Predose (0-4 Hr), 0.5, 4, 24, 72Hr post Cy1 D1 dose (infusion duration=1.5 Hr); Day 8 of Cy 1, 2, 4; predose, 0.5 Hr postose on Day 1 of Cy2, 3, 4, 6, every 4 Cy thereafter (up to Cy16); study completion/ET (approximately 6.75 years) (Cy=14 days)
Half-Life (t1/2) of MEHD7945A | Predose (0-4 Hr), 0.5, 4, 24, 72Hr post Cy1 D1 dose (infusion duration=1.5 Hr); Day 8 of Cy 1, 2, 4; predose, 0.5 Hr postose on Day 1 of Cy2, 3, 4, 6, every 4 Cy thereafter (up to Cy16); study completion/ET (approximately 6.75 years) (Cy=14 days)
Accumulation Ratio of MEHD7945A | Predose (0-4 Hr), 0.5, 4, 24, 72Hr post Cy1 D1 dose (infusion duration=1.5 Hr); Day 8 of Cy 1, 2, 4; predose, 0.5 Hr postose on Day 1 of Cy2, 3, 4, 6, every 4 Cy thereafter (up to Cy16); study completion/ET (approximately 6.75 years) (Cy=14 days)
Recommended Phase 2 Dose (RP2D) of MEHD7945A | Days 1-28
Percentage of Participants With an Objective Response (Complete Response [CR] or Partial Response [PR]) Assessed by the Investigator Using Response Evaluation Criteria in Solid Tumors Version 1.0 (RECIST V1.0) | From the first study treatment (Cy1 D1, 1 Cy=14 days) to first occurrence of progression or death within 60 days of the last administration of study drug, whichever occurs first (up to approximately 6.75 years)
Duration of Objective Response (CR or PR) Assessed by the Investigator Using Response Evaluation Criteria in Solid Tumors Version 1.0 (RECIST V1.0) | First occurrence of a documented objective response until the time of relapse or death within 60 days of the last administration of study drug, whichever occurs first (up to approximately 6.75 years)
Progression-Free Survival (PFS) Assessed by the Investigator Using Response Evaluation Criteria in Solid Tumors Version 1.0 (RECIST V1.0) | From the first study treatment (Cy1 D1, 1 Cy = 14 days) to first occurrence of progression or death within 60 days of the last administration of study drug, whichever occurs first (up to approximately 6.75 years)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Pirzkall, M.D., Study Director — Genentech, Inc.
Locations (6):
- United States (3):
  - Uni of Colorado Cancer Center; Anschutz Cancer Pavilion, Aurora, Colorado
  - Massachusetts General Hospital., Boston, Massachusetts
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas
- Spain (3):
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - HOSPITAL DE MADRID NORTE SANCHINARRO- CENTRO INTEGRAL ONCOLOGICO CLARA CAMPAL; Servicio de Oncologia, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia